CLINICAL TRIAL: NCT01678287
Title: A Phase 1, Double-Blind, Placebo-Controlled, Randomized Study to Assess the Pharmacokinetics, Safety and Tolerability of Repeat Oral Dosing of ASP1941 and to Explore the Effect of ASP1941 on Glucose Levels in Healthy Adult Subjects (18 to 45 Years and ≥ 65 Years)
Brief Title: Study of the Pharmacokinetics of ASP1941 and the Effect on Glucose Concentrations in Male and Female Young and Elderly Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 1941-CL-0052
Record Dates: First submitted 2012-08-27; First posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Healthy Volunteers; Pharmacokinetics of ASP1941
Keywords: ASP1941
MeSH Terms: interventions — ipragliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 Non elderly receiving ASP1941 (Experimental): healthy subjects age 18 to 45 years receiving ASP1941
  Interventions: Drug: ASP1941
- Arm 2 Non elderly receiving placebo (Experimental): healthy subjects age 18 to 45 years receiving placebo
  Interventions: Drug: Placebo
- Arm 3 Elderly receiving ASP1941 (Experimental): healthy subjects age ≥ 65 years receiving ASP1941
  Interventions: Drug: ASP1941
- Arm 4 Elderly receiving placebo (Experimental): healthy subjects age ≥ 65 years receiving placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP1941 — oral
  Arms: Arm 1 Non elderly receiving ASP1941; Arm 3 Elderly receiving ASP1941
Drug: Placebo — oral
  Arms: Arm 2 Non elderly receiving placebo; Arm 4 Elderly receiving placebo

SUMMARY:
This is a study of the pharmacokinetic profile and safety and tolerability of ASP1941after repeat dosing and the effect of ASP1941 on glucose levels in non elderly and elderly healthy adult male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, healthy non-elderly (age 18-45 years, inclusive) or healthy elderly (age 65 or over)
* If female, subject is not pregnant or nursing, and uses medically acceptable contraceptive method to prevent pregnancy from screening until study discharge
* Body weigh between 60 and 100kg and body Mass Index between 20 and 30kg/m2, inclusive
* Negative urine screen for drugs of abuse, including alcohol and cotinine

Exclusion Criteria:

* History of type 1 or type 2 diabetes
* Fasting plasma glucose level higher than 6.4mmol/L or hemoglobin A1c level higher than 6.2%
* Presence of renal glucosuria and/or proteinuria
* Clinically significant history of asthma, eczema, and or any other allergic condition.
* Clinically significant history of upper gastrointestinal symptoms within the 4 weeks prior to admission to the clinical unit.
* History of any clinically significant neurological, gastrointestinal, renal, hepatic, pulmonary, metabolic, cardiovascular, psychiatric, endocrine, hematological disorder or disease, or any other medical condition that would preclude participation in the study.
* History of multiple drug allergies or a known allergy or suspected hypersensitivity to the study drug or any chemically related derivatives of the study drug or any components of the formulation
* Has hepatitis or a positive result to serology test for hepatitis A antibody Immunoglobulin M, hepatitis B surface antigen or hepatitis C virus at screening
* Known to be positive for human immunodeficiency virus antibodies.
* Donated one unit (450 mL) or more of blood or plasma within 60 days prior to the first dose of study medication.
* Has a history of consuming more than an average of 2 ounces of alcohol-containing products per day or a history of alcoholism or drug/chemical abuse within the last 3 years.
* Use of any tobacco or nicotine-containing products within 120 days prior to the first dose of study medication.
* Taken any prescribed systemic or topical medication within 21 days prior to the first dose of study medication with the exception of contraceptives to prevent pregnancy.
* Taken any systemic or topical over-the counter medication, complementary or alternative medications, e.g., vitamins, herbal, or nutritional supplements, with the exception of acetaminophen, within 10 days prior to the first dose of study medication.
* Taken an investigational drug within 30 days of the first dose of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AEs) | Through Day 29
Safety as assessed by vital signs, electrocardiogram (ECG), physical examination, and laboratory evaluations | Through Day 29
Pharmacokinetic profile of ASP1941 (plasma):AUCtau, CL/F, Cmax, tmax, t1/2, Vz/F, PTR | Days 1 and 18 pre-dose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
  Area under the curve over the time interval between consecutive dosing (AUCtau),Apparent total body clearance after extravascular dosing (CL/F), Maximum observed concentration (Cmax), Time to reach Cmax (Tmax), Terminal elimination half-life (t1/2), Apparent volume of distribution during the terminal phase after single or repeated extravascular dosing (Vz/F), Peak Trough Ratio (PTR)
Pharmacokinetic profile of ASP1941 (urine): Ae, Ae%, Aelast, Aelast%, Ae24, CLR | Day 1 at pre-dose and from 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, 48 to 72, 72 to 96 hours post-dose
  Cumulative amount of drug excreted into urine up to the ending time of the last collection period (Ae), Fraction of the drug excreted in urine (Ae) in % up to the ending time of last collection period (Ae%), Cumulative amount of drug or glucose excreted into urine up to the collection time of the last measurable amount (Aelast),Fraction of drug excreted into urine (Ae) in % up to the collection time of the last measurable concentration (Aelast% ), Fraction of glucose excreted into urine up to 24 hrs (Ae24), Renal clearance (CLR)
Pharmacokinetic profile of ASP1941 (urine): Aetau, Aetau%, Aelast, CLR | Day 18 at pre-dose and from 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12, 12 to 24, 24 to 36, 36 to 48, 48 to 72, 72 to 96 hours post-dose
  Cumulative amount of drug or glucose excreted into urine over the time interval between consecutive dosing (Aetau ), Fraction of drug or glucose excreted into urine (Aetau) in % over the time interval between consecutive dosing (Aetau%)

SECONDARY OUTCOMES:
Pharmacodynamic profile of blood glucose: Cmax and AUCtau | Day -1 at -24, -23.75, -23.5, -23, -22.5, -22, -21, -20, -18, -16, -12, -8 and 0 (predose) hours prior to dose on Day 1 and on Day 18 predose and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post-dose
Pharmacodynamic profile of urine glucose: Aelast and Aetau | Day 1 and Day 18
Rate of glucose excretion per sampling interval | Day 1 and Day 18
Rate of glucose excretion over 24 hours | Day 1 and Day 18

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Comprehensive Phase One, Miramar, Florida, United States